CLINICAL TRIAL: NCT04878302
Title: Improving Symptom Trajectories of Tic Disorders and Co-occurring Diagnoses: The Role of Integrative Intensive Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-20-0562
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Tic Disorder, Childhood; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Tic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Eligible families will be randomly assigned to an immediate treatment group or a 1-month waitlist.
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators assessing outcomes are kept unaware of the specific treatment condition and pre-treatment assessment scores.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Taming Tics Together Protocol (Experimental): Families will participate in the 5-day telehealth-based intensive intervention and will receive three treatment formats which will provide CBIT and co-occurring diagnosis treatment:
  1. Child/teen-only groups
  2. Individual one-to-one sessions
  3. Parent/caregiver-only groups
  Interventions: Behavioral: Combination of Comprehensive Behavioral Intervention for Tics (CBIT) and Evidence-based interventions for co-occurring diagnoses (i.e., Cognitive Behavioral Therapy, Behavioral Parent Training)
- 1-Month Waitlist Control (No Intervention): Families in the 1-month waitlist control group will participate in the initial intake assessment, then receive no treatment for a 1-month period. Following the 1-month period, families will participate in an assessment, then will be offered a place in a Taming Tics Together group

INTERVENTIONS:
Behavioral: Combination of Comprehensive Behavioral Intervention for Tics (CBIT) and Evidence-based interventions for co-occurring diagnoses (i.e., Cognitive Behavioral Therapy, Behavioral Parent Training) — Families assigned to the immediate treatment group will receive the telehealth-based Taming Tics Together protocol(created using well-established, evidence-based treatment protocols), which includes group (parent/caregiver-only, child/teen-only) and individualized one-to-one sessions to address tics and co-occurring diagnoses.
  Arms: Experimental: Taming Tics Together Protocol

SUMMARY:
The purpose to the current study was to examine the efficacy of a telehealth, group-based, combined and intensive intervention for youth with tic disorders (TDs) and common co-occurring diagnoses. Families seeking treatment for TDs and common co-occurring diagnoses will be randomly assigned to receive treatment immediate (enrollment in the next group) or remain on a 1-month waitlist, and then receive treatment. Outcomes will be assessed across the treatment phase, immediately following treatment (post), as well as 1-month following the end of treatment.

DETAILED DESCRIPTION:
Over 1,000,000 children in the U.S. have a tic disorder (TD). TDs can substantially impact daily child functioning across numerous domains leading to a significant public health impact of TDs. Additionally, an overwhelming majority of children with a TD have at least one co-occurring disorder. Over 60% also meet criteria for attention deficit/hyperactivity disorder (ADHD), half struggle with anxiety and at least a third have clinically elevated Obsessive Compulsive-spectrum symptoms.

Comprehensive Behavioral Intervention for Tics (CBIT) is a first-line treatment for youth with TDs. It has been shown to be effective in reducing the frequency, duration, and severity of tics in children and adolescents. Nonetheless, access to trained CBIT providers remains limited, and common comorbid conditions are not addressed in standard CBIT. Thus, there is a desperate need for interventions that can simultaneously increase CBIT access and incorporate treatment strategies for comorbidities.

Intensive, group-based interventions are well-established for the treatment of comorbid disorders and have been shown to be a cost-efficient modality for delivering multimodal interventions. Intensive formats provide the opportunity for families to gain access to treatment for a limited time without the extended burden often associated with weekly treatment sessions. Further, intensive group-based treatments can simultaneously treat comorbidities.

To address the critical need for increasing access to CBIT and simultaneously treating common comorbidities, a week-long group-based intensive intervention for children with TDs and common co-occurring diagnoses (Taming Tics Together) has been developed and will be evaluated. Participants will be randomly assigned to immediate treatment or a 1-month waitlist control. Assessments will take place pre-treatment, daily throughout the intervention, as well as at 1-month post treatment.

The primary aims of the current study are to evaluate symptom reduction in tic severity and co-occurring condition symptom severity. Importantly, the investigators seek to learn more about the effectiveness of an intensive-format for tics and co-occurring diagnoses, which may lead to mechanisms to improve access to care for families who often are not able to access effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Youth participants are between seven and 17 years old
* Meet diagnostic criteria for a primary or co-primary diagnosis of a Tic Disorder
* Are available to participate in all sessions
* Are comfortable in English
* Youth participants have at least borderline clinician symptoms of ADHD, oppositional defiant disorder (ODD), obsessive compulsive disorder (OCD) and/or an anxiety disorder.

Exclusion Criteria:

* Are identified as having a psychiatric condition that is more impairing and requiring treatment prior to a tic intervention.
* Meet criteria for Autism Spectrum Disorder.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | Change from pre-treatment to post, and 1-month following the end of treatment
  Yale Global Tic Severity Scale (Leckman et al., 1989). The Yale Global Tic Severity Scale is a clinician-administered assessment evaluating tic history, as well as tics present over the past 7-10 days. The Yale Global Tic Severity Scale has been used in several randomized controlled trials and has exhibited excellent internal consistency (i.e., McGuire et al., 2018). Motor and vocal tics are rated based on their number, frequency, intensity, complexity and interference (each rated on a scale from 0-5), and impairment (rated on a scale from 0-50). The Total Tic Severity Score evaluates overall motor and vocal tic severity (range 0-50), and the Total Yale Global Tic Severity Scale Score evaluates the total tic severity score in additional to impairment, with a range of scores from 0 to 100. Higher scores indicate increased severity.

SECONDARY OUTCOMES:
Revised Child Anxiety and Depression Scale (RCADS) | Change from pre-treatment to post and 1-month
  Revised Child Anxiety and Depression Scale (RCADS; Chorpita et al., 2000). The RCADS is a 47-item self-report measure to evaluate several internalizing domains. Items are rated on a scale from 0 (never) to 3 (always). The RCADS has demonstrated high internal consistency (Chorpita, Moffit, & Gray, 2005)).
Disruptive Behavior Disorder Rating Scale (DBD-RS) | Change from pre-treatment to post and 1-month following the end of treatment.
  Disruptive Behavior Disorder Rating Scale (DBD-RS; Pelham et al.,1992). The DBD-RS is a 45-item parent rating scale to assess for disruptive behaviors, specifically, ADHD, oppositional defiant disorder, and conduct disorder. Informants complete the rating scale using a four-point Likert scale (zero = not at all; one = just a little; two = pretty much; three = very much). The DBD-RS has demonstrated high internal consistency (Pelletier et al., 2006).

CONTACTS AND LOCATIONS:
Locations (1):
- Florida International University, Miami, Florida, United States

REFERENCES:
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] Pelham WE Jr, Gnagy EM, Greenslade KE, Milich R. Teacher ratings of DSM-III-R symptoms for the disruptive behavior disorders. J Am Acad Child Adolesc Psychiatry. 1992 Mar;31(2):210-8. doi: 10.1097/00004583-199203000-00006. PMID 1564021
- [Background] Pelletier, J, Collett, B, Gimpel, G, & Crowley S. Assessment of Disruptive Behaviors in Preschoolers: Psychometric Properties of the Disruptive Behavior Disorders Rating Scale and School Situations Questionnaire. Journal of Psychoeducational Assessment. 2006; 24(1): 3-18.
- [Background] Chorpita BF, Moffitt CE, Gray J. Psychometric properties of the Revised Child Anxiety and Depression Scale in a clinical sample. Behav Res Ther. 2005 Mar;43(3):309-22. doi: 10.1016/j.brat.2004.02.004. PMID 15680928
- [Background] Chorpita BF, Yim L, Moffitt C, Umemoto LA, Francis SE. Assessment of symptoms of DSM-IV anxiety and depression in children: a revised child anxiety and depression scale. Behav Res Ther. 2000 Aug;38(8):835-55. doi: 10.1016/s0005-7967(99)00130-8. PMID 10937431
- [Background] Woods, D, Piacentini, J, Chang, S, Deckersbach, T, Ginsburg, G, Peterson, A, Scahill, L, Walkup, J, & Wilhelm, S. Managing Tourette Syndrome: A Behavioral Intervention for Children and Adults Therapist Guide. 2008; New York, NY: Oxford University Press.
- [Background] McGuire JF, Piacentini J, Storch EA, Murphy TK, Ricketts EJ, Woods DW, Walkup JW, Peterson AL, Wilhelm S, Lewin AB, McCracken JT, Leckman JF, Scahill L. A multicenter examination and strategic revisions of the Yale Global Tic Severity Scale. Neurology. 2018 May 8;90(19):e1711-e1719. doi: 10.1212/WNL.0000000000005474. Epub 2018 Apr 13. PMID 29653992